CLINICAL TRIAL: NCT01231009
Title: The Role of Corticosteroids and Vestibular Exercises in Recovery of Vestibular Neuritis: a Prospective Randomized Controlled Clinical Trial
Brief Title: The Role of Corticosteroids and Vestibular Exercises in Recovery of Vestibular Neuritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: 1st ENT Department, AHEPA University Hospital, John Goudakos, Research fellow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VN-01-JG
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-01

CONDITIONS: Vestibular Neuritis
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroids (Active Comparator): Patients receive for 7 days intravenous corticosteroids, dexamethasone, and they continue receiving for 7 days corticosteroids per os
  Interventions: Drug: Corticosteroids; Other: Vestibular exercises
- Vestibular exercises (Placebo Comparator): Patients perform for 15 days certain vestibular exercises under suspicion of an expert physiotherapist
  Interventions: Drug: Corticosteroids; Other: Vestibular exercises

INTERVENTIONS:
Drug: Corticosteroids — Intravenous Dexamethasone, 8mg three times per day tapering down for 7 days Per os dexamethasone, 2mg per day tapering down for 7 days
Other: Vestibular exercises — Vestibular exercises in order to enhance vestibulo-ocular reflex for 15 days under the suspicion of physiotherapist

SUMMARY:
Aim of present study is to determine whether corticosteroids and vestibular exercises are equal effective in the recovery of balance in patients with acute vestibular neuritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of acute or sub-acute rotatory vertigo with postural imbalance, nausea and imbalance.
* Horizontal-rotatory spontaneous nystagmus.

Exclusion Criteria:

* History of vestibular disfunction before the acute onset of symptoms
* Simultaneous Hearing loss
* Neurologic disorder
* Pregnancy or lactation
* History of psychiatric disorders
* History of glaucoma
* Diabetes
* Hypertension
* Contraindication in receiving corticosteroids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
clinical recovery of vestibular function | 1 year
  clinical examination (nystagmus, Romberg test, head-thrust test, head-shaking test) and questionnaires (Greek edition of Dizziness Handicap Inventory and European Evaluation of Vertigo Scale)
Laboratory recovery of vestibular | 1 year
  caloric test and vestibular evoked myogenic potentials

CONTACTS AND LOCATIONS:
Locations (1):
- 1st ENT Department, AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Derived] Goudakos JK, Markou KD, Psillas G, Vital V, Tsaligopoulos M. Corticosteroids and vestibular exercises in vestibular neuritis. Single-blind randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2014 May;140(5):434-40. doi: 10.1001/jamaoto.2014.48. PMID 24604142